CLINICAL TRIAL: NCT06633783
Title: A Multicenter, Randomized, Open-label, Parallel-controlled Phase III Study Comparing the Efficacy and Safety of Semaglutide Injection and Wegovy® for Weight Loss in Obese Subjects
Brief Title: A Phase III Study Comparing the Weight Loss Effects of Semaglutide Injection and Wegovy®
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hangzhou Jiuyuan Gene Engineering Co. Ltd., (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JY29-2-302
Record Dates: First submitted 2024-10-07; First posted 2024-10-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-06

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — semaglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Semaglutide injection (Experimental): Semaglutide：0.25 mg、0.5 mg、1.0mg、1.7mg、2.4mg
  Interventions: Drug: Semaglutide
- Wegovy® (Active Comparator): Wegovy®：0.25 mg、0.5 mg、1.0mg、1.7mg、2.4mg
  Interventions: Drug: Semaglutide

INTERVENTIONS:
Drug: Semaglutide — The dose escalation phase, starting with 0.25mg once weekly and increasing every 4 weeks (0.5mg, 1.0mg, 1.7mg), is expected to last 16 weeks; In the dose maintenance phase, the target dose of 2.4mg was maintained for 28 weeks.Treatment duration 44 weeks.
  Arms: Semaglutide injection
Drug: Semaglutide — The dose escalation phase, starting with 0.25mg once weekly and increasing every 4 weeks (0.5mg, 1.0mg, 1.7mg), is expected to last 16 weeks; In the dose maintenance phase, the target dose of 2.4mg was maintained for 28 weeks.Treatment duration 44 weeks.
  Arms: Wegovy®

SUMMARY:
The purpose of the study is to compare the effect on body weight in subjects taking semaglutide injection or subjects taking Wegovy®.

DETAILED DESCRIPTION:
The study will involve participants engaging in discussions with study staff regarding healthy dietary choices, strategies for increasing physical activity, and additional methods for achieving weight loss, alongside the administration of the study medication. Participants will be randomly assigned to receive either semaglutide injection or Wegovy®. The study medication will be administered via a weekly subcutaneous injection using a fine needle in the abdominal skinfold. The duration of the study will be approximately 2 years, during which participants will attend 13 clinic visits with the study physician.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily participate in this trial and sign the informed consent form.
2. Male or female, aged 18-75 years (inclusive) at the time of signing the informed consent form.
3. Body mass index (BMI) ≥28.0 kg/m2 at screening. （4）At least one self-reported unsuccessful weight loss history.

Exclusion Criteria:

* Blood Glucose-Related:

  1. Glycated hemoglobin (HbA1c) level ≥6.5% at screening.
  2. History of type 1 or type 2 diabetes.
  3. Received hypoglycemic drug treatment within 90 days prior to screening.
  4. Received GLP-1 receptor agonist treatment within 180 days prior to screening.
* Obesity-Related:

  （5）Self-reported weight change >5 kg within 90 days prior to screening, regardless of medical history.

  （6）Received any drug treatment for obesity within 90 days prior to screening. （7）Previous or planned surgical or device treatment for obesity during the trial period, except for the following: (1) liposuction and/or abdominal lipolysis performed >1 year prior to screening; (2) gastric banding with the band removed >1 year prior to screening; (3) intragastric balloon placement with the balloon removed >1 year prior to screening.
* Psychological Health-Related:

  （8）History of severe depression or a Patient Health Questionnaire-9 (PHQ-9) score ≥15 at screening.

  （9）Diagnosed with other severe mental illnesses, including schizophrenia, schizoaffective disorder, paranoid psychosis, bipolar (affective) disorder, epilepsy-induced mental disorder, and mental retardation with mental disorders.

  （10）History of suicidal behavior. （11）Suicidal ideation corresponding to type 4 or 5 on the Columbia-Suicide Severity Rating Scale (C-SSRS) at screening.
* General Safety:

  （12） Thyroid diseases: Including a personal or family history of medullary thyroid carcinoma (MTC) or multiple endocrine neoplasia type 2 (MEN2); or calcitonin (CT) ≥50ng/L at screening; or thyroid-stimulating hormone (TSH) >6.0mIU/L or <0.4mIU/L at screening; or concurrent hyperthyroidism.

  (13) History of acute or chronic pancreatitis, or blood amylase ≥3×ULN at screening, or triglycerides (TG) ≥5.65 mmol/L (500 mg/dL) at screening.

  (14) Alanine aminotransferase (ALT) ≥3×ULN, aspartate aminotransferase (AST) ≥3×ULN, or total bilirubin (TBiL) ≥3×ULN at screening.

  (15) Serum creatinine level ≥1.5 mg/dL (132μmol/L) in males or ≥1.4 mg/dL (123μmol/L) in females at screening.

  (16) Untreated or poorly controlled hypertension (defined as systolic blood pressure ≥160 mmHg and/or diastolic blood pressure ≥100 mmHg).

  (17) Severe cardiac history, defined as New York Heart Association (NYHA) class III and IV at screening, and/or hospitalization for unstable angina pectoris or transient ischemic attack within 60 days prior to screening, and/or stroke (except lacunar infarction) or myocardial infarction within 180 days prior to screening.

  (18) Gastrointestinal diseases assessed by the investigator to potentially increase the risk after medication (such as obstructive diseases: pyloric obstruction and intestinal obstruction; or gastrointestinal motility disorders: postoperative gastroparesis, idiopathic gastroparesis; or severe active ulcers, etc.).

  (19) Known or suspected allergy to any component of semaglutide injection or other GLP-1 receptor agonists.

  (20) Use of drugs that may cause significant weight gain within 90 days prior to screening or expected during the trial, including systemic glucocorticoid therapy for more than 1 week; tricyclic antidepressants (such as amitriptyline, imipramine, clomipramine, doxepin); antipsychotic or antiepileptic drugs (such as mirtazapine, paroxetine, phenelzine, chlorpromazine hydrochloride, chlorpromazine, olanzapine, valproic acid and its derivatives, lithium preparations, methimazole).

  (21) Obesity caused by other endocrine diseases, including hypothalamic obesity, pituitary obesity, hypothyroid obesity, Cushing's syndrome, insulinoma, acromegaly, pseudohypoparathyroidism, and hypogonadism.

  (22) Known subjects planned for hospitalization for any surgical treatment during the trial at screening.

  (23) Participated in other clinical trials and used investigational drugs within 90 days prior to screening.

  (24) History of drug abuse (including drug addiction) and/or alcohol dependence within 180 days prior to screening.

  (25) Diagnosed with malignant tumors within 5 years prior to screening (except for adequately treated cervical carcinoma in situ, basal cell or squamous cell skin cancer, local prostate cancer after radical surgery, and breast ductal carcinoma in situ after radical surgery).

  (26) Pregnant or lactating women, females or males with reproductive plans during the trial period or unwilling to use effective contraceptive methods.

  (27) Subjects who, in the investigator's judgment, have any disease or other conditions that may endanger their safety or affect their compliance with the protocol, making them unsuitable for participation in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 370 (Estimated)
Dates: Start 2024-10-30 (Estimated); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Change in body weight | From baseline at week 0 to week 44
  Percent

SECONDARY OUTCOMES:
Change in body weight | From baseline at week 0 to week 28
  Percent
Subjects who achieve body weight reduction equal to or above 5% | From baseline at week 0 to week 44
  Number of subjects
Subjects who achieve body weight reduction equal to or above 10% | From baseline at week 0 to week 44
  Number of subjects
Subjects who achieve body weight reduction equal to or above 15% | From baseline at week 0 to week 44
  Number of subjects
Change in body mass index (BMI) | From baseline at week 0 to week 44
  kg/m^2
Change in waist circumference | From baseline at week 0 to week 44
  cm
Change in systolic blood pressure and diastolic blood pressure | From baseline at week 0 to week 44
  mmHg
Change in lipids | From baseline at week 0 to week 44
  mg/dL

CONTACTS AND LOCATIONS:
Locations (14):
- China (14):
  - Xuancheng People's Hospital, Xuancheng, Anhui
  - Huizhou Central People's Hospital, Huizhou, Guangdong
  - Luoyang Third People's Hospital, Luoyang, Henan
  - The First Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan
  - The First Affiliated Hospital of Nanyang Medical College, Nanyang, Henan
  - The Second Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Yichang Central People's Hospital, Yichang, Hubei
  - Huai an First People's Hospital, Huaian, Jiangsu
  - The Second People's Hospital of Lianyungang, Lianyungang, Jiangsu
  - The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Affiliated Hospital of Jiangsu University, Zhenjiang, Jiangsu
  - Central Hospital Affiliated to Shandong First Medical University, Jinan, Shandong
  - Jincheng Grand Hospital, Jincheng, Shanxi

IPD SHARING:
Plan to Share IPD: No